CLINICAL TRIAL: NCT02647788
Title: Pilot Study, Blinded Randomized Control Trial, Single Center Study to Compare Acetaminophen & Codeine Versus Ibuprofen/Acetaminophen for Pain Control and Patient Satisfaction After Ambulatory Hand Surgery
Brief Title: Acetaminophen/Codeine vs Acetaminophen/Ibuprofen for Pain Control and Patient Satisfaction After Hand Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BACH-2015, 823043
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Pain, Postoperative
Keywords: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Ibuprofen; acetaminophen, codeine drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetaminophen/Ibuprofen (Active Comparator): Group 1: Acetaminophen 650 mg; Ibuprofen 400 mg
  Interventions: Drug: Acetaminophen/Ibuprofen
- Acetaminophen/Codeine (Active Comparator): Group 2: Acetaminophen 300mg, Codeine 30 mg
  Interventions: Drug: Acetaminophen/Codeine

INTERVENTIONS:
Drug: Acetaminophen/Ibuprofen — After hand surgery, take Acetaminophen 650 mg/Ibuprofen 400 mg every 6 hours as needed for pain until postoperative clinic visit
  Other Names: Tylenol/Advil
  Arms: Acetaminophen/Ibuprofen
Drug: Acetaminophen/Codeine — After hand surgery, take Acetaminophen 300mg/Codeine 30 mg every 6 hours as needed for pain until postoperative clinic visit
  Other Names: Tylenol 3
  Arms: Acetaminophen/Codeine

SUMMARY:
The purpose of this research study is to find out if taking Acetaminophen with Ibuprofen (e.g. Tylenol + Advil), a non-opioid regimen, provides the same type of pain relief after hand surgery compared to Acetaminophen and codeine (e.g. Tylenol 3), an opioid regimen.

DETAILED DESCRIPTION:
Primary Objective:

To establish, through a randomized control trial, whether post-operative Acetaminophen and Ibuprofen (non-opioid regimen) would provide equivalent post-operative analgesia to ambulatory hand surgery patients compared to Acetaminophen and Codeine (opioid regimen).

Secondary Objective:

To establish whether the opioid versus non-opioid post-operative pain regimen influences patient satisfaction.

Sixty-three patients enrolled for each group (non-opioid and opioid). Approximately 145 patients will be required to achieve complete data for 63 patients in each group (assuming 15% lost to follow-up & failure to comply with study protocol).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ambulatory hand surgery for carpal tunnel and trigger finger, under local anesthesia with or without sedation.

Exclusion Criteria:

* ASA> 3;
* Coagulopathy;
* Renal disease,
* Liver disease,
* History of recent gastro-intestinal bleeding
* Pregnancy.
* Diagnosis of chronic pain currently taking opioid pain medication or with a history of drug abuse.
* Patients with a self-described allergy to ASA, acetaminophen, NSAIDS and codeine.
* All patients receiving a brachial plexus block for anesthesia and/or analgesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2015-12; Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Steinberg, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited between 11/18/15 and 1/10/18 and were identified on the physicians surgery schedule as patients receiving either trigger finger or carpel tunnel surgery.
Pre-assignment Details: There were 4 patients that were enrolled but did not make it to the randomization stage. 2 patients had liver disease and therefore met exclusion criteria for the study. The other 2 patients did not have surgery.
Period: Overall Study
Arm/Group | Acetaminophen/Ibuprofen | Acetaminophen/Codeine
Started | 70 | 70
Completed | 54 | 57
Not Completed | 16 | 13
Not completed — Lost to Follow-up | 13 | 11
Not completed — Did not want opiate | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Felt itchy with assigned medication | 1 | 0
Not completed — Felt nauseous with assigned medication | 1 | 1

BASELINE CHARACTERISTICS:
Population: 144 patients were consented for this study. There were 4 patients that were enrolled but did not make it to the randomization stage and 140 patients were placed into the study. 111 patients completed the study and were included in analysis.
Groups:
- Acetaminophen/Ibuprofen: Group 1: Acetaminophen 650 mg; Ibuprofen 400 mg
  Acetaminophen/Ibuprofen: After surgery, take Acetaminophen 650 mg/Ibuprofen 400 mg every 6 hours as needed for pain until postoperative clinic visit
- Acetaminophen/Codeine: Group 2: Acetaminophen 300mg, Codeine 30 mg
  Acetaminophen/Codeine: After surgery, take Acetaminophen 300mg/Codeine 30 mg every 6 hours as needed for pain until postoperative clinic visit
- Total: Total of all reporting groups
Arm/Group | Acetaminophen/Ibuprofen | Acetaminophen/Codeine | Total
Number analyzed (Participants) | 54 | 57 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (12) | 59 (13) | 59 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 17 | 19 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 19 | 36
  White | 32 | 36 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
VAS Pain Score [Mean (Standard Deviation); unit: units on a scale] — The visual analog scale (VAS) for pain is a patient reported outcome measurement. It is a continuous scale anchored by no pain (0) and worst pain imaginable (10).
  units on a scale | 1.93 (2.04) | 2.50 (2.51) | 2.22 (2.30)

OUTCOME MEASURES:

1. Primary Outcome: Assessing Change in Pain Using the Visual Analogue Scale (VAS) Pain Score
Description: To establish, through a randomized control trial, whether post-operative Acetaminophen and Ibuprofen (non-opioid regimen) would provide equivalent post-operative analgesia to ambulatory hand surgery patients compared to Acetaminophen and Codeine (opioid regimen). The pain VAS is a continuous scale where 0=no pain and 10=worst pain imaginable.
Time Frame: Subjects reported pain 3 times a day each day after hand surgery (at dinner time, before going to sleep and in the middle of the night), until post-op appointment (between 4 and 8 days after surgery). The numbers reported are the average daily pain scores
Population: 111 patients completed the study and their data was included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acetaminophen/Ibuprofen | Acetaminophen/Codeine
Number analyzed (Participants) | 54 | 57
score on a scale
  VAS Pain Day 1: number analyzed (Participants) | 49 | 53
  VAS Pain Day 1 | 2.90 (2.22) | 3.51 (2.69)
  VAS Pain Day 2: number analyzed (Participants) | 43 | 47
  VAS Pain Day 2 | 2.36 (2.31) | 2.40 (2.52)
  VAS Pain Day 3: number analyzed (Participants) | 37 | 40
  VAS Pain Day 3 | 1.69 (2.00) | 2.26 (2.38)
  VAS Pain Day 4: number analyzed (Participants) | 35 | 35
  VAS Pain Day 4 | 1.47 (1.82) | 1.93 (2.01)
  VAS Pain Day 5: number analyzed (Participants) | 30 | 34
  VAS Pain Day 5 | 1.23 (1.61) | 1.48 (1.48)
  VAS Pain Day 6: number analyzed (Participants) | 29 | 30
  VAS Pain Day 6 | 1.29 (1.49) | 1.35 (1.37)
  VAS Pain Day 7: number analyzed (Participants) | 23 | 27
  VAS Pain Day 7 | 1.17 (1.38) | 1.01 (1.21)

2. Secondary Outcome: Quality of Recovery-9 (QoR-9).
Description: To establish whether the opioid versus non-opioid post-operative pain regimen influences patient satisfaction through Quality of Recovery (QoR) scores in ambulatory hand surgery. This 9 question survey has a maximum score (best outcome) of 18 and minimum (worst outcome) of 3. The survey was administered over the phone on post-operative day 2.
Time Frame: Postoperative Day 2
Population: Of the 111 subjects that completed the study, QoR score was available for 93 participants.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Acetaminophen/Ibuprofen | Acetaminophen/Codeine
Number analyzed (Participants) | 44 | 49
Scores on a scale | 16.91 (1.38) | 16.65 (1.91)

3. Secondary Outcome: Number of Pills Used
Time Frame: From the time of surgery to first clinic visit (post-op day 6 to 8)
Population: Of the 111 subjects that completed the study, data about how many capsules were used was available for 100 participants.
Measure: Mean (Standard Deviation); unit: Pills
Arm/Group | Acetaminophen/Ibuprofen | Acetaminophen/Codeine
Number analyzed (Participants) | 50 | 50
Pills | 13.72 (8.04) | 14.14 (9.77)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the subjects time participating on the study. Participation began on the subject's surgery day and ended at their first clinical visit (6-8 days after surgery).
Arm/Group | Acetaminophen/Ibuprofen | Acetaminophen/Codeine
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 32/70 | 30/70
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acetaminophen/Ibuprofen (N=70) | Acetaminophen/Codeine (N=70)
Nausea (General disorders) | 8 | 7
Constipation (General disorders) | 8 | 12
Itchiness (General disorders) | 12 | 11
Dizziness (General disorders) | 3 | 2
Drowsiness (General disorders) | 22 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT02647788/Prot_SAP_000.pdf